CLINICAL TRIAL: NCT04338178
Title: Efficacy of a Multi-component Treatment Program Integrating Cognitive - Affective - Addictive Based Intervention in Obese Patients: a Prospective Multicentric Randomized Clinical Trial
Brief Title: Efficacy of a Cognitive - Affective - Addictive Based Intervention to Decrease Food Craving in Obese Patients.
Acronym: OBESADEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHUBX 2017/50
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Craving; Cognitive Behavioral Therapy; Cognitive Remediation Therapy; Addiction
MeSH Terms: conditions — Obesity; Behavior, Addictive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Standard outpatient program, with additional group sessions integrating the experimental intervention : Cognitive Remediation Therapy (CRT), Emotional Skills Training (EST), and Cognitive Behavioral Therapy focused on craving and food addiction (CBT), delivered once a week during 10 weeks.
  Interventions: Behavioral: Cognitive Remediation Therapy (CRT); Behavioral: Emotional Skills Training (EST); Behavioral: Cognitive Behavioral Therapy
- Standard intervention (Active Comparator): Standard outpatient program, with additional group sessions integrating control intervention : multidisciplinary outpatient program including several consultations with endocrinologists, dietitians, psychologists, nutritionists and/or physical activity coaches, delivered once a week during 10 weeks.
  Interventions: Procedure: Multidisciplinary outpatient program

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy (CRT) — This intervention consists of mental exercises aimed at improving executive function via practice. Simple cognitive tasks that encourage reflective learning and insight into patient's own thinking process are administered. Exercises target set-shifting (i.e., cognitive flexibility), estimating, organization and planning.
  Arms: Experimental intervention
Behavioral: Emotional Skills Training (EST) — EST places emphasis on the improvement of inner emotion awareness, facial and body expression recognition and intra- and interpersonal emotion regulation skills. Different modules and interactive exercises are designed to help patients learn about i) the functions and manifestations of emotions, ii) the identification and labelling of own's and others' emotions, iii) tolerating and communicating emotions, and iiii) balancing between negative and positive emotions.
  Arms: Experimental intervention
Behavioral: Cognitive Behavioral Therapy — CBT intervention aimed to manage food craving by teaching group members cognitive (e.g., restructuring of urge-related thoughts) and behavioural strategies (e.g., increasing awareness through food diaries, relaxation skills, identification of cues that trigger craving, avoidance of high-risk situations for craving, distraction).
  Arms: Experimental intervention
Procedure: Multidisciplinary outpatient program — Multidisciplinary outpatient program including several consultations with endocrinologists, dietitians, psychologists, nutritionists and/or physical activity coaches. Patients are regularly followed and educated about the importance of lifestyle changes including healthy dietary habits and exercise in weight reduction and maintenance. Patients are also usually given information about nutritional value of various foods and few simple exercises for decreasing and maintaining body weight. This program is therefore planned as part of the usual care and responds to the recommendations of good practice for obesity
  Arms: Standard intervention

SUMMARY:
Since the 80's, the prevalence of obesity has more than doubled and despite progression of knowledge, interventions usually lead to a transient reduction in body weight that is not maintained in the long-term. These failures in weight management may be partly explained by an incomplete understanding of obesity risk and maintaining factors.

Behavioral and neurobiological similarities between use of high palatable foods and addictive psychoactive drugs have led to the concept of food addiction. Addiction is defined as a loss of control of use, and its persistence despite accumulation of negative consequences. Craving, an uncontrollable and involuntary urge to use, has shown to be a core determinant of persistent use and relapse in addiction. Recent studies have established that food addiction, craving and emotional eating concern a large part of obese patients, and that food addiction may explain some negative outcomes of weight loss treatments, such as unsuccessful attempts to reduce calories and early termination of treatment programs.

Recent advances in neuropsychiatry suggest that an imbalanced interplay between cognitive and affective processes impedes self-control and enhances over- or under-controlled behaviors. In the field of food intake and weight management, there is increasing evidence that besides environmental factors, inefficient executive functions and emotion regulation skills are salient phenomena underlying habit-forming processes that are present in eating disorder subtypes as well as obesity. This has led some authors to consider disordered eating behaviors as 'allostatic' reactions by which the modulation of food intake is used by vulnerable individuals to adjust to craving, maladaptive cognitive and/or emotional strategies.

Current recommendations emphasize the need for translating these discoveries into treatments to promote healthy eating and weight management.

Over the last 5 years, a growing base of clinical and behavioural studies have indicated that, individually, Cognitive-Behavioural Therapy (CBT), Emotional Skills Training (EST), and Cognitive Remediation Therapy (CRT) are promising techniques to decrease disordered eating behaviors, including craving.

The investigators hypothesize that addition to treatment as usual (TAU) of a specific program targeting executive functions, emotional regulation, and addictive-like eating behaviors, could have a beneficial impact on reported food craving, and improve weight management among obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Treatment seeking obese patients (30 kg/m2 ≤ BMI ≤ 45 kg/m2)
* Report at least one food craving episode in the 30 days before pre-inclusion visit (assessed by one question adapted from the State version of the Food Cravings Questionnaire, FCQ-S)
* Able to participate in group sessions once a week for 10 weeks
* Affiliated person or beneficiary of a social security scheme

Exclusion Criteria:

* Severely impaired physical and/or mental health that, according to the investigator, may affect the participant's compliance with the study and understanding of assessment tools
* Difficulty in understanding and / or writing French
* Hypothalamic obesity
* Impossibility to be reached by telephone
* Individuals participating in another study that includes an ongoing exclusion period
* Be deprived of liberty due to an ongoing legal procedure
* Pregnancy or breastfeeding
* Individuals under legal protection or unable to express personally their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Food Cravings Questionnaire-Trait-reduced (FCQ-T-r) score | Baseline (T0) and 12 weeks (T1)
  Self-administered questionnaire consisting of 15 items assessing several aspects of food craving: lack of control over eating, thoughts or preoccupation with food, intentions and plans to consume food, emotions before or during food craving, cues that may trigger food craving

SECONDARY OUTCOMES:
Body mass index (BMI) | 12 weeks (T1)
  Body mass index (BMI) is a measure of body fat based on height and weight, expressed in kg/m2
Body mass index (BMI) | 6 months (T2)
  Body mass index (BMI) is a measure of body fat based on height and weight, expressed in kg/m2
Waist circumference | 12 weeks (T1)
  Waist circumference measured following the WHO STEPwise approach to surveillance (STEPS) and their corresponding guidelines for physical measurement
Waist circumference | 6 months (T2)
  Waist circumference measured following the WHO STEPwise approach to surveillance (STEPS) and their corresponding guidelines for physical measurement
Percentage of body fat and fat-free mass | 12 weeks (T1)
  Bio Impedance Analysis (BIA) is a more specific measure of body composition and adiposity. The variables of interest will be the percentages of body fat and fat-free mass.
Percentage of body fat and fat-free mass | 6 months (T2)
  Bio Impedance Analysis (BIA) is a more specific measure of body composition and adiposity. The variables of interest will be the percentages of body fat and fat-free mass.
Emotional Appetite Questionnaire (EMAQ) Score | 12 weeks (T1)
  Emotional Appetite Questionnaire (EMAQ) contains 22 items assessing variations of food intake in response to emotional states and situations. 9 items evaluate negative emotions, 5 evaluate positive emotions, 5 refer to negative situations and 3 to positive situations.A score is calculated for positive emotions (EMAQ-PE), negative emotions (EMAQ-NE), positive situations (EMAQ-PS) and negative situations (EMAQ-NS). For each subscale, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. A positive total score (EMAQ-P) is obtained by averaging the EMAQ-PE and EMAQ-PS scores. A negative total score (EMAQ-N) is obtained by averaging the EMAQ-NE and EMAQ.
Emotional Appetite Questionnaire (EMAQ) Score | 6 months (T2)
  Emotional Appetite Questionnaire (EMAQ) contains 22 items assessing variations of food intake in response to emotional states and situations. 9 items evaluate negative emotions, 5 evaluate positive emotions, 5 refer to negative situations and 3 to positive situations.A score is calculated for positive emotions (EMAQ-PE), negative emotions (EMAQ-NE), positive situations (EMAQ-PS) and negative situations (EMAQ-NS). For each subscale, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. A positive total score (EMAQ-P) is obtained by averaging the EMAQ-PE and EMAQ-PS scores. A negative total score (EMAQ-N) is obtained by averaging the EMAQ-NE and EMAQ.
Eating Disorder Examination-Questionnaire (EDE-Q) Score | 12 weeks (T1)
  Eating Disorder Examination-Questionnaire (EDE-Q) includes 36-item assessing the frequency of disordered eating behaviors over the past 28 days. The EDE-Q provides subscale scores reflecting the severity of aspects of the psychopathology of eating disorders. The subscales are Restraint, Eating Concern, Shape Concern and Weight Concern. To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. If ratings are only available on some items, a score may nevertheless be obtained by dividing the resulting total by the number of rated items as long as more than half the items have been rated. To obtain total score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e. four). The variables of interest will be the EDE-Q total score and subscales' scores.
Eating Disorder Examination-Questionnaire (EDE-Q) Score | 6 months (T2)
  Eating Disorder Examination-Questionnaire (EDE-Q) includes 36-item assessing the frequency of disordered eating behaviors over the past 28 days. The EDE-Q provides subscale scores reflecting the severity of aspects of the psychopathology of eating disorders. The subscales are Restraint, Eating Concern, Shape Concern and Weight Concern. To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. If ratings are only available on some items, a score may nevertheless be obtained by dividing the resulting total by the number of rated items as long as more than half the items have been rated. To obtain total score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e. four). The variables of interest will be the EDE-Q total score and subscales' scores.
Dutch Eating Behaviour Questionnaire (DEBQ) Score | 12 weeks (T1)
  Dutch Eating Behaviour Questionnaire (DEBQ) consists of 33 items and assesses on a 5-point Likert scale, ranging from "never" to "very often" external, restraint and emotional eating. For the study, only the 10 items of the external eating subscale will be used. The variable of interest will be the corresponding External eating subscale score.
Dutch Eating Behaviour Questionnaire (DEBQ) Score | 6 months (T2)
  Dutch Eating Behaviour Questionnaire (DEBQ) consists of 33 items and assesses on a 5-point Likert scale, ranging from "never" to "very often" external, restraint and emotional eating. For the study, only the 10 items of the external eating subscale will be used. The variable of interest will be the corresponding External eating subscale score.
modified Yale Food Addiction Scale (mYFAS) Assessment | 12 weeks (T1)
  modified Yale Food Addiction Scale (mYFAS) 2.0 : is a 35-item self-report scale assessing Food Addiction (FA) symptoms based on the 11 diagnostic criteria for substance related and addictive disorders proposed in the DSM-5. FA is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress. The variables of interest will be the number of symptoms and the presence (vs absence) of a FA diagnosis.
modified Yale Food Addiction Scale (mYFAS) Assessment | 6 months (T2)
  modified Yale Food Addiction Scale (mYFAS) 2.0 : is a 35-item self-report scale assessing Food Addiction (FA) symptoms based on the 11 diagnostic criteria for substance related and addictive disorders proposed in the DSM-5. FA is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress. The variables of interest will be the number of symptoms and the presence (vs absence) of a FA diagnosis.
Psychiatric disorders assessment using the Mini International Neuropsychiatric Interview (MINI) | 6 months (T2)
  Mini International Neuropsychiatric Interview (MINI) is a structured diagnostic interview providing standardized assessment of psychiatric disorders defined according to Axis I DSM-5 : eating disorders, addictive disorders, mood disorders, anxiety disorders, and attention deficit hyperactivity disorder The variables of interest will be the proportion of patients with each of types of disorders. The number of comorbid psychiatric conditions will also be assessed using four categories : no comorbid disorder, one comorbid disorder, two comorbid disorders, three or more comorbid disorders
Interviewer Severity Rating (ISR) established for Addiction Severity Index (ASI) | 6 months (T2)
  Addiction Severity Index (ASI) : is a semi-structured interview to assess impairments that commonly occur due to substance-related disorders . It explores seven areas that may be affected by addiction: medical status, employment/support status, substance and behavioral addiction, family and social relationships, legal status, and psychological status. For each area explored, an Interviewer Severity Rating (ISR) is established, from 0 to 9, reflecting the severity in the considered area. A score equal or above 4 reflects a need for additional treatment. ASI ISRs will be dichotomized to less than 4 or 4 and more (important need for additional treatment). The variables of interest will be the proportion of patients with need for additional treatment in each of the seven areas
Trail Making Test (TMT) completion time and number of perseverative errors | 12 weeks (T1)
  Trail Making Test (TMT) : is used to measure cognitive and motor speed and mental flexibility. The variables of interest will the difference in completion time between TMT B and TMT A (TMT B - TMT A) and the number of perseverative errors on the TMT B.
Wisconsin Card Sorting Test 64 (WCST) number and percentage of perseverative errors | 12 weeks (T1)
  Wisconsin Card Sorting Test 64 (WCST) : measures categorisation, inference, testing of hypotheses, cognitive flexibility, cognitive inhibition and response to feedback. The variable of interest will be the number and percentage of perseverative errors
Zoo test Score | 12 weeks (T1)
  Zoo test : Is a subtest of the Behavioural Assessment of the Dysexecutive Syndrome (BADS). It provides information about subjects' ability to plan a route to visit six of a possible 12 locations in a zoo, firstly in a demanding, open-ended situation where little external structure is provided, and secondly in a situation that involves simply following a concrete, externally imposed strategy. The map and rules have been constructed so that there are only four variations on a route through the zoo that can be followed in order that none of the rules of the test are infringed. There are two trials. A profile score is computed based on planning time, execution time and the number of errors for both trials. The maximum profile score is of 4. The variable of interest will be the total profile score
UPPS Impulsive Behavior Scale Score | 12 weeks (T1)
  The UPPS Impulsive Behavior Scale evaluates in 20 items five different impulsivity facets (4 items each) : Negative Urgency, Positive Urgency, Lack of Premeditation, Lack of Perseverance and Sensation Seeking. Each item are rated on Likert scale ranging from 1 ("I agree strongly") to 4 (" I disagree strongly"). For each subscale, a mean score of the available items is calculated. The variables of interest will be the five different impulsivity facets scores
Monetary Choice Questionnaire (MCQ) | 12 weeks (T1)
  Monetary Choice Questionnaire (MCQ) includes a fixed set of 27 items with immediate rewards ranging from $11-$78 and delayed rewards ranging from $25-$85 with a delay of 7-186 days. Delayed rewards are grouped into three categories based on size, with nine items per category. Participants' hyperbolic discount parameter (k value) is determined by fitting data a discount function equation. The variables of interest will be the k value and the proportion of participants by k rank
Performances (flexibility) at the Stroop and Verbal Fluency computerized tests (EMA). | 12 weeks (T1)
  Total number of correct words serves as the primary performance score
Difficulties in Emotion Regulation Scale (DERS) Score | 12 weeks (T1)
  Difficulties in Emotion Regulation Scale (DERS) is a 36-item measure that assesses individuals' typical levels of difficulties in emotion regulation with six subscale: (a) nonacceptance of emotional responses, (b) difficulty engaging in goal-directed behavior when distressed, (c) impulse control difficulties when distressed, (d) lack of awareness of emotions, (e) limited access to strategies for regulation, and (f) lack of emotional clarity. For each subscale, a score is calculated by summing responses from relevant items. A total score is obtained by adding each subscale score. The variable of interest will be the DERS total score
Difficulties in Emotion Regulation Scale (DERS) Score | 6 months (T2)
  Difficulties in Emotion Regulation Scale (DERS) is a 36-item measure that assesses individuals' typical levels of difficulties in emotion regulation with six subscale: (a) nonacceptance of emotional responses, (b) difficulty engaging in goal-directed behavior when distressed, (c) impulse control difficulties when distressed, (d) lack of awareness of emotions, (e) limited access to strategies for regulation, and (f) lack of emotional clarity. For each subscale, a score is calculated by summing responses from relevant items. A total score is obtained by adding each subscale score. The variable of interest will be the DERS total score
Depression Anxiety Stress Scales (DASS-21) Score | 12 weeks (T1)
  Depression Anxiety Stress Scales (DASS-21) : is a 21-item measure of negative emotional symptoms that evaluates three dimensions: depression, anxiety and stress (7 items per subscale). A 4-point severity scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), measures the extent to which each emotional state has been experienced over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. Scores obtained will need to be multiplied by 2 to calculate the final score of each dimension. The variables of interest will be the three dimensions' scores.
Depression Anxiety Stress Scales (DASS-21) Score | 6 months (T2)
  Depression Anxiety Stress Scales (DASS-21) : is a 21-item measure of negative emotional symptoms that evaluates three dimensions: depression, anxiety and stress (7 items per subscale). A 4-point severity scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), measures the extent to which each emotional state has been experienced over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. Scores obtained will need to be multiplied by 2 to calculate the final score of each dimension. The variables of interest will be the three dimensions' scores.
Quality Of Life, Obesity and Dietetics rating scale (QOLOD) Score | 12 weeks (T1)
  Quality Of Life, Obesity and Dietetics rating scale (QOLOD) includes 36 items designed to assess quality of life in 5 domains: physical impact, psycho-social impact, impact on sex life , comfort with food, and diet experience The variables of interest will be the 5 subscales scores
Quality Of Life, Obesity and Dietetics rating scale (QOLOD) Score | 6 months (T2)
  Quality Of Life, Obesity and Dietetics rating scale (QOLOD) includes 36 items designed to assess quality of life in 5 domains: physical impact, psycho-social impact, impact on sex life , comfort with food, and diet experience The variables of interest will be the 5 subscales scores
Number of sessions completed (Compliance) | After the 10th session (S10)
  Compliance at group session will correspond to the number of sessions completed out of the 10 proposed group sessions.
Patient Satisfaction Questionnaire (PSQ) Score | After the 3rd session (Week 3)
  Patient Satisfaction Questionnaire (PSQ) includes 6 domains of satisfaction that are rated on a 10-points Likert scale as well as 2 open questions on what was helpful and what could be improved. For both groups (i.e experimental intervention and control intervention), the variable of interest will be the a mean total score of satisfaction in each of the 6 domains. In addition, for the group receiving the experimental intervention, scores of satisfaction in each of the 6 domains will be described separately for the CRT, EST and CBT modules of the intervention
Patient Satisfaction Questionnaire (PSQ) Score | After the 6th session (Week 6)
  Patient Satisfaction Questionnaire (PSQ) includes 6 domains of satisfaction that are rated on a 10-points Likert scale as well as 2 open questions on what was helpful and what could be improved. For both groups (i.e experimental intervention and control intervention), the variable of interest will be the a mean total score of satisfaction in each of the 6 domains. In addition, for the group receiving the experimental intervention, scores of satisfaction in each of the 6 domains will be described separately for the CRT, EST and CBT modules of the intervention
Patient Satisfaction Questionnaire (PSQ) Score | After the 9th session (Week 9)
  Patient Satisfaction Questionnaire (PSQ) includes 6 domains of satisfaction that are rated on a 10-points Likert scale as well as 2 open questions on what was helpful and what could be improved. For both groups (i.e experimental intervention and control intervention), the variable of interest will be the a mean total score of satisfaction in each of the 6 domains. In addition, for the group receiving the experimental intervention, scores of satisfaction in each of the 6 domains will be described separately for the CRT, EST and CBT modules of the intervention
Motivation to change Score | 12 weeks (T1)
  Motivation to change will be assessed explore beliefs about the importance to change and perceived ability to change. Rating scores are based on a Likert 0-10 scale. Higher scores indicate more positive beliefs about one's importance/ability to change. These two scores will be used as variables of interest
Revised Helping Alliance Questionnaire (HAQ-11) Score | 12 weeks (T1)
  Revised Helping Alliance Questionnaire (HAQ-11) is a 11-item questionnaire that measures the strength of the patient-therapist therapeutic alliance. A total score is obtained by summing the item scores. The variable of interest will be the HAQ-11total score
Ecological Momentary Assessment data collection | During 7 days after baseline
  will be acquired by 5 signal-based assessments per day. One random assessment Ecological Momentary Assessment data collection will occur during each of the following time periods: 9:00 am to 11:00 am; 11:00 am to 2:00 pm; 2:00 pm to 5:00 pm; 5:00 pm to 8:00 pm; and 8:00 pm to 10:00 pm during 7 days. The questions administered after random prompt will include items relative to eating behaviors, craving and food intake, exposure to food cues, positive and negative affectivity, the experience of stress (type of stress and level of perceived stress), other personal states, cognitive functioning, craving and emotional regulation strategies.
Ecological Momentary Assessment data collection | During 7 days after the 10th session (Week 10 to week 11)
  will be acquired by 5 signal-based assessments per day. One random assessment Ecological Momentary Assessment data collection will occur during each of the following time periods: 9:00 am to 11:00 am; 11:00 am to 2:00 pm; 2:00 pm to 5:00 pm; 5:00 pm to 8:00 pm; and 8:00 pm to 10:00 pm during 7 days. The questions administered after random prompt will include items relative to eating behaviors, craving and food intake, exposure to food cues, positive and negative affectivity, the experience of stress (type of stress and level of perceived stress), other personal states, cognitive functioning, craving and emotional regulation strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Mélina FATSEAS, Principal Investigator — University Hospital, Bordeaux; Sylvie BERTHOZ, Study Director — CNRS UMR 5287 - INCIA
Locations (3):
- France (3):
  - Assistance Publique Hôpitaux de Paris Hôpital Européen Georges Pompidou, Paris
  - Assistance Publique Hôpitaux de Paris Hôpital Ambroise Paré, Paris
  - CHU de Bordeaux, Pessac

IPD SHARING:
Plan to Share IPD: Undecided